CLINICAL TRIAL: NCT02023840
Title: The Use of Erythritol Powder and Locally Derived Metronidazole for the Non-surgical Treatment of Periodontitis: a Split-mouth Randomized Controlled Clinical Trial
Brief Title: The Use of Erythritol Powder and Metronidazole Gel for the Non-surgical Treatment of Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Proed, Torino, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07.2013.ERYTHRITOL.PROED
Record Dates: First submitted 2013-12-18; First posted 2013-12-30 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: Periodontal Pocket
Keywords: periodontitis; pockets
MeSH Terms: conditions — Periodontal Pocket; Periodontitis | interventions — High-Energy Shock Waves; Erythritol

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrasonics and erythritol, metronidazole gel (Active Comparator): Scaling and root planing with ultrasonics and erythritol air powder will be followed by application of metronidazole gel
  Interventions: Drug: metronidazole gel; Procedure: ultrasonics; Procedure: erythritol
- ultrasonics and erythritol, placebo (Placebo Comparator): Scaling and root planing with ultrasonics and erythritol air powder will be followed by application of placebo
  Interventions: Procedure: ultrasonics; Procedure: erythritol; Drug: placebo

INTERVENTIONS:
Drug: metronidazole gel
  Arms: ultrasonics and erythritol, metronidazole gel
Procedure: ultrasonics
Procedure: erythritol
Drug: placebo
  Arms: ultrasonics and erythritol, placebo

SUMMARY:
Aim of the present study is evaluate the use of erythritol powder with/without the adjunct of local metronidazole in the treatment of periodontal pockets.

20 consecutive adult periodontal patients, requiring cause-related therapy as phase 1 of their treatment plan, and presenting ≥4 sites with probing pocket depth ≥4mm will be enrolled. For each patients four sites will be considered for the study, and two sites will be allocated in the test group and two sites will be allocated in the control group. In the test group, ultrasonic debridement of the pocket will be performed using a piezoceramic ultrasonic device with the a tip connected to the handpiece for 5 minutes/pocket. Then, it will be followed by the subgingival use of erythritol powder 2x5 seconds/pocket. At this time the subgingival delivery of metronidazole gel will be provided. In the control group, the same protocol will be used except for the use of a placebo instead of metronidazole. After instrumentation, patients will rinse with chlorhexidine 0.20% 3 times/day for 2 weeks.

At baseline, 1 month, 3 months and 6 months the following parameters will be evaluated: Probing Pocket depth (PPD), Bleeding on Probing (BoP), Clinical Attachment Level (CAL).

DETAILED DESCRIPTION:
The long term results and benefit of infection control in the treatment of periodontal disease have been well documented. According to a cause-related concept, the disruption of bacterial plaque biofilms can be defined as primary objective for the treatment of periodontitis.

In the past few years, glycine powder air polishing showed positive outcomes in removing subgingival biofilm in periodontal pockets, and subgingivally delivered metronidazole seemed to improve the results of scaling and root-planing alone . Recently, a new prophylactic powder has been developed. The special action of the powder is attributable to the new ingredient Erythritol and the extra-fine grains that measure only 14 microns. The small size results on one hand in a minimal impact per grain on the treated surface and on the other hand in a very dense jet of powder, efficient on biofilm.

Aim of the present study is evaluate the use of erythritol powder with/without the adjunct of local metronidazole in the treatment of periodontal pockets.

MATERIALS & METHODS:

20 consecutive adult periodontal patients, requiring cause-related therapy as phase 1 of their treatment plan, and presenting ≥4 sites with probing pocket depth ≥4mm will be enrolled. For each patients four sites will be considered for the study, and two sites will be allocated in the test group and two sites will be allocated in the control group. In the test group, ultrasonic debridement of the pocket will be performed using a piezoceramic ultrasonic device with the tip connected to the Handpiece Led for 5 minutes/pocket. Then, it will be followed by the subgingival use of erythritol powder applied by the use of Perio-Flow Handpiece with Perio-Flow Nozzle, connected to an airflow unit 2x5 seconds/pocket. At this time the subgingival delivery of metronidazole gel will be provided. In the control group, the same protocol will be used except for the use of a placebo instead of metronidazole. After instrumentation, patients will rinse with chlorhexidine 0.20% 3 times/day for 2 weeks.

At baseline, 1 month, 3 months and 6 months the following parameters will be evaluated: Probing Pocket depth (PPD), Bleeding on Probing (BoP), Clinical Attachment Level (CAL).

ELIGIBILITY:
Inclusion Criteria:

* adult patients suffering from periodontitis at least 4 sites with probing pocket depth =>4mm

Exclusion Criteria:

* Heavy smokers current pregnant patients history of malignancy Long term steroidal or antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Probing pocket Depth change | baseline, 6 months
  Using a periodontal calibrated PCP-15 mm probe, the pocket depth will be measured
Bleeding on Probing change | baseline, 6 months
  Using a periodontal calibrated PCP-15 mm probe, the bleeding on probing will be detected
Clinical Attachment level change | baseline, 6 months
  Using a periodontal calibrated PCP-15 mm probe, the attachment level will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Cardaropoli, DDS, Principal Investigator — Proed, Torino, Italy
Locations (1):
- PROED, Institute for Professional Education in Dentistry, Torino, Italy

IPD SHARING:
Plan to Share IPD: No